CLINICAL TRIAL: NCT00827905
Title: Remote Doppler System to Measure Heart Rate and Breathing Pattern
Brief Title: Substantial Equivalence Study for Kai Sensors RSpot Non-Contact Respiratory Rate Spot Check
Status: Completed | Type: Observational
Sponsor: Kai Medical, Inc. (Industry)
Responsible Party: Amy Droitcour, Director of Technology, Kai Medical, Inc.
Other Study IDs: KAI-00003; RA-2008-061
Record Dates: First submitted 2009-01-21; First posted 2009-01-23 (Estimated); Last update posted 2010-08-06 (Estimated); Status verified 2010-08

CONDITIONS: Respiration
Keywords: Non-Contact; Radar; Respiratory; Respiration; Breathing; Rate; Frequency; Respiratory Mechanics; Respiratory Rate Measurement
MeSH Terms: conditions — Respiratory Aspiration

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Hospitalized: Patients admitted to the hospital
  Interventions: Device: RSpot Non-Contact Respiratory Rate Spot Check

INTERVENTIONS:
Device: RSpot Non-Contact Respiratory Rate Spot Check — The Kai Sensors RSpot 100 provides a measurement of respiratory rate at a single point in time. It uses a low-power radar to detect respiratory effort, and analyzes the respiratory effort signal to provide a respiratory rate.
  Other Names: KaiSpot; RSpot 100; RSpot; Non-Contact Respiratory Rate Spot Check

SUMMARY:
The purpose of this study is to determine whether the respiratory rate provided by the Kai Sensors RSpot 100 Non-Contact Respiratory Rate Spot Check is as accurate as that provided by the Welch Allyn Propaq Encore model 242 and the Embla Embletta system with Universal XactTrace respiratory effort sensor and Somnologica for Embletta software.

DETAILED DESCRIPTION:
Currently, medical professionals obtain respiratory rate for vital signs assessments either by counting the number of breaths during a 15, 30, or 60 second interval and multiplying to obtain breaths per minute, or by reading the respiratory rate off of a multiparameter vital signs monitor (such as a Welch Allyn Propaq Monitor), that provides respiratory effort information based on the change of AC impedance through ECG leads. The Respiration channel (RESP) of the Welch Allyn Propaq is intended to detect the rate or absence of respiratory effort, deriving the signal by measuring the AC impedance between the selected terminals of the ECG electrodes. The RSpot 100 Non-Contact Respiratory Rate Spot Check provides an alternative to the medical professional counting respiratory rate or reading the rate from a vital signs monitor designed for continuous respiratory rate monitoring. The Kai Sensors RSpot 100 Non-Contact Respiratory Rate Spot Check is used for a one-time measurement of respiratory rate as part of a vital signs assessment in the hospital or other clinical settings.

In this study, the RSpot is operated simultaneously with two other systems that provide a respiratory rate: Welch Allyn Propaq Encore model 242 and Embletta system with Universal XactTrace and Somnologica software. A respiratory rate is also obtained by counting respiratory excursions for the same duration as the RSpot measurement interval, 15, 30, or 60 seconds. The rates obtained from each of the four measurement methods are then compared.

ELIGIBILITY:
Inclusion Criteria:

* Adult >18 years old
* Hospitalized on Tower 6 or Pauahi 6 or Pauahi 4
* Clinically stable
* Able to provide informed consent

Exclusion Criteria:

* Clinically unstable

  1. Hypotensive requiring pressors or intra-aortic balloon pump
  2. Intubated
  3. Dyspnea or chest pain at rest
  4. Resting tachycardia (heart rate >100 bpm)
  5. Requires supplemental (e.g., nasal canula or face mask) oxygen
* Scheduled or planned (e.g., CT scan, central line placement) procedure during the 30 minute study period

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients Hospitalized at the Queen's Medical Center in Honolulu, HI
Sampling Method: Non-Probability Sample
Enrollment: 20 (Estimated)
Dates: Start 2009-01; Primary Completion 2009-01 (Actual); Study Completion 2009-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Todd Seto, MD, Principal Investigator — The Queen's Medical Center; Olga Boric-Lubecke, PhD, Study Director — University of Hawaii
Locations (1):
- The Queen's Medical Center, Honolulu, Hawaii, United States